CLINICAL TRIAL: NCT06735547
Title: Effectiveness of a Mobile Telerehabilitation Tool Versus Conventional Treatment in Total Knee Arthroplasty: a Controlled Clinical Trial
Brief Title: Effectiveness of a Mobile Telerehabilitation Tool Versus Conventional Treatment in Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanitas University (Other)
Collaborators: Biokeralty Research Institute (Industry)
Responsible Party: Principal Investigator, Claudia Aristizábal, Director research unit, Sanitas University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 102-22UNV
Record Dates: First submitted 2024-11-18; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-10

CONDITIONS: Musculoskeletal Disorders; Knee Osteoarthritis (OA)
Keywords: Knee replacement arthroplasty; Telerehabilitation; Mobile applications; Artificial intelligence; Outpatient management
MeSH Terms: conditions — Musculoskeletal Diseases; Osteoarthritis, Knee | interventions — Telerehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- Telerehabilitation (Experimental): Patients will receive telerehabilitation by means of the TRAK mobile tool, collecting data and allowing them to monitor their activity through ROM during exercises (bio-feedback).
  Interventions: Device: Telerehabilitation
- Conventional Therapy (Active Comparator): Patients will be assessed by a professional physiotherapist, who will monitor their progress, by measuring range of motion (ROM), and stability, making corrections if necessary.
  Interventions: Other: Conventional therapy group

INTERVENTIONS:
Device: Telerehabilitation — Patients in the Telerehabilitation group will perform an average of three therapy sessions per week, with data collected and monitored by TRAK's physiotherapists. Both groups will have their results measured monthly by the orthopedic surgeons for 12 weeks (3 months) postoperatively.
  Arms: Telerehabilitation
Other: Conventional therapy group — Patients in the conventional group will be assessed by a professional physiotherapist, scheduling appointments according to their own preferences and disponibility. Both groups will have their results measured monthly by the orthopedic surgeons for 12 weeks (3 months) postoperatively.
  Arms: Conventional Therapy

SUMMARY:
Knee arthroplasty is one of the most common surgical procedures, and early rehabilitation is essential for patient recovery, pain modulation and a faster reintegration into daily life activities. However, it has been reported that the percentage of patients who continue rehabilitation for the time required to achieve these outcomes is much lower than those who abandon therapy. This is often due to various factors such as office hours, difficult access to appointments, and sometimes insufficient infrastructure and personnel to meet the demand. Currently, due to the global situation, it is crucial to conduct these rehabilitation processes remotely and virtually, making use of various technological tools that enable patients to interact with the healthcare professionals in charge of their rehabilitation. Among these tools are mobile applications on smartphones, which not only facilitate proper physical preparation, but also offer valuable real-time feedback. Furthermore, 8% of the total cost of knee joint replacements corresponds to the rehabilitation program. These costs are significantly reduced with telerehabilitation assisted by mobile tools, which not only improves patient access but also increases adherence and satisfaction levels by allowing the customization of rehabilitation programs based on each patient's specific needs and characteristics. The aim of this study is to evaluate the effectiveness outcomes of an artificial intelligence-guided mobile tool versus conventional rehabilitation during the first three months postoperatively following total knee replacement.

DETAILED DESCRIPTION:
A parallel, controlled randomized clinical trial will be conducted. Study Population: Patients with knee osteoarthritis undergoing primary total knee replacement (TKR) at Clínica Universitaria Colombia and Puente Aranda Emergency Center, whose postoperative follow-up is ambulatory, and who meets the inclusion criteria.

Outcomes: Functionality will be the primary outcome, measured in terms of the WOMAC score, knee range of movement, and pain, by means of the visual analogue scale. Adherence to treatment, number of therapy sessions, patient satisfaction, and the presence of adverse events will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with degenerative osteoarthritis with an indication for primary Total Knee Replacement (TKR) surgery at Clínica Universitaria Colombia or Central de Urgencias de Puente Aranda.
* Patients in the postoperative period following primary outpatient TKR.
* Patients with functional independence.
* Patients who agree to participate in the study and sign the informed consent form.
* Patients with access to a mobile device, tablet, computer, with internet access and the ability to operate it.
* Patients who have an appropriate space to perform therapy at home.
* Patients who will be accompanied during therapy sessions at home.

Exclusion Criteria:

* ASA Class IV (American Society of Anesthesiologists)
* BMI > 35
* Dementia and cognitive impairment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Knee Range of Motion | Measurement will be performed before surgery (at the preoperative visit) and monthly during the first three months of the postoperative period (ending at 3 months postoperatively).
  Measurement of knee joint range of motion in flexion and extension using a goniometer from preoperative follow-up to the third month postoperatively.
Functionality - WOMAC survey | Measurement will be performed before surgery (at the preoperative visit) and monthly during the first three months of the postoperative period (ending at 3 months postoperatively).
  WOMAC survey, validated in Colombia with a numerical result from 0 to 96, carried out during the preoperative visit until the third postoperative month.
Functionality - Get Up and Go | Measurement will be performed before surgery (at the preoperative visit) and monthly during the first three months of the postoperative period (ending at 3 months postoperatively).
  Test that measures the time required to get up from the chair, walk to the mark 3 meters away, turn around and sit back in the chair, measured from preoperative follow-up to the third month postoperatively.
Pain - Visual Analogue Scale | Measured from day 0 every 24 hours until day 14 postoperatively.
  Measurement of the patient's subjective perception of pain in a written survey and scale from 0 to 10.

SECONDARY OUTCOMES:
Number of therapy sessions | From the beginning of rehabilitation until the third postoperative month.
  Number of face-to-face physical therapy sessions or TRAK therapy sessions.
Percentage of Adherence | From the beginning of rehabilitation until the third postoperative month.
  Percentage of adherence to the prescribed rehabilitation program.
Patient Satisfaction | Measured at the end of rehabilitation, 3 months postoperatively
  Measuring patient satisfaction with the prescribed rehabilitation program through a question with the option to respond: completely satisfied, satisfied, neither satisfied nor dissatisfied, somewhat satisfied, and not at all satisfied
Surgery Complications | Measured from the start of surgery to the third month postoperatively.
  Complications derived from the surgical procedure: Material Failure, Dislocation, Fracture, Wound Dehiscence, Rigidity, Readmission, Death, Need for mobilization under anesthesia
Therapy Adverse Events | Measured from the start of the postoperative period to the third postoperative month.
  Adverse events that occurred during the prescribed therapy sessions: Fall, Wound Dehiscence, Fracture, Ecchymosis, Ligament Injury, Need for intervention, Hematoma, Other

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica Universitaria Colombia, Bogotá, Bogota D.C., Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pellegrini CA, Lee J, DeVivo KE, Harpine CE, Del Gaizo DJ, Wilcox S. Reducing sedentary time using an innovative mHealth intervention among patients with total knee replacement: Rationale and study protocol. Contemp Clin Trials Commun. 2021 Jun 18;22:100810. doi: 10.1016/j.conctc.2021.100810. eCollection 2021 Jun. PMID 34195473
- [Background] Eichler S, Rabe S, Salzwedel A, Muller S, Stoll J, Tilgner N, John M, Wegscheider K, Mayer F, Voller H; ReMove-It study group. Effectiveness of an interactive telerehabilitation system with home-based exercise training in patients after total hip or knee replacement: study protocol for a multicenter, superiority, no-blinded randomized controlled trial. Trials. 2017 Sep 21;18(1):438. doi: 10.1186/s13063-017-2173-3. PMID 28934966
- [Background] Khan F, Ng L, Gonzalez S, Hale T, Turner-Stokes L. Multidisciplinary rehabilitation programmes following joint replacement at the hip and knee in chronic arthropathy. Cochrane Database Syst Rev. 2008 Apr 16;2008(2):CD004957. doi: 10.1002/14651858.CD004957.pub3. PMID 18425906
- [Background] Muller M, Toussaint R, Kohlmann T. [Total hip and knee arthroplasty : Results of outpatient orthopedic rehabilitation]. Orthopade. 2015 Mar;44(3):203-11. doi: 10.1007/s00132-014-3000-0. German. PMID 25209014
- [Background] Callejas-Cuervo M, Gutierrez RM, Hernandez AI. Joint amplitude MEMS based measurement platform for low cost and high accessibility telerehabilitation: Elbow case study. J Bodyw Mov Ther. 2017 Jul;21(3):574-581. doi: 10.1016/j.jbmt.2016.08.016. Epub 2016 Sep 9. PMID 28750967
- [Background] van Egmond MA, van der Schaaf M, Vredeveld T, Vollenbroek-Hutten MMR, van Berge Henegouwen MI, Klinkenbijl JHG, Engelbert RHH. Effectiveness of physiotherapy with telerehabilitation in surgical patients: a systematic review and meta-analysis. Physiotherapy. 2018 Sep;104(3):277-298. doi: 10.1016/j.physio.2018.04.004. Epub 2018 Jun 19. PMID 30030037
- [Background] Backer HC, Wu CH, Schulz MRG, Weber-Spickschen TS, Perka C, Hardt S. App-based rehabilitation program after total knee arthroplasty: a randomized controlled trial. Arch Orthop Trauma Surg. 2021 Sep;141(9):1575-1582. doi: 10.1007/s00402-021-03789-0. Epub 2021 Feb 6. PMID 33547927
- [Background] Tripuraneni KR, Foran JRH, Munson NR, Racca NE, Carothers JT. A Smartwatch Paired With A Mobile Application Provides Postoperative Self-Directed Rehabilitation Without Compromising Total Knee Arthroplasty Outcomes: A Randomized Controlled Trial. J Arthroplasty. 2021 Dec;36(12):3888-3893. doi: 10.1016/j.arth.2021.08.007. Epub 2021 Aug 9. PMID 34462184
- [Background] Henderson KG, Wallis JA, Snowdon DA. Active physiotherapy interventions following total knee arthroplasty in the hospital and inpatient rehabilitation settings: a systematic review and meta-analysis. Physiotherapy. 2018 Mar;104(1):25-35. doi: 10.1016/j.physio.2017.01.002. Epub 2017 Feb 1. PMID 28802773
- [Background] Masaracchio M, Hanney WJ, Liu X, Kolber M, Kirker K. Timing of rehabilitation on length of stay and cost in patients with hip or knee joint arthroplasty: A systematic review with meta-analysis. PLoS One. 2017 Jun 2;12(6):e0178295. doi: 10.1371/journal.pone.0178295. eCollection 2017. PMID 28575058
- [Background] Hsu H, Siwiec RM. Knee Osteoarthritis. StatPearls. Treasure Island (FL). 2024. Available from: https://www.ncbi.nlm.nih.gov/books/NBK507884/
- [Background] Jiang S, Xiang J, Gao X, Guo K, Liu B. The comparison of telerehabilitation and face-to-face rehabilitation after total knee arthroplasty: A systematic review and meta-analysis. J Telemed Telecare. 2018 May;24(4):257-262. doi: 10.1177/1357633X16686748. Epub 2016 Dec 27. PMID 28027679